CLINICAL TRIAL: NCT03344419
Title: Glutamatergic Modulation to Facilitate the Behavioral Treatment of Cocaine Use Disorders
Status: Suspended | Phase: Phase 3 | Type: Interventional
Why Stopped: Funding
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Elias Dakwar, research psychiatrist, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 7461; 5U01DA040647-04 (NIH)
Record Dates: First submitted 2017-11-13; First posted 2017-11-17 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Cocaine Use Disorder
Keywords: cocaine; mindfulness based relapse prevention; motivational enhancement therapy
MeSH Terms: interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CI-581a+MET+MBRP (Experimental): Administration of CI-581a at 0.71 mg/kg during weeks 1 and 5 combined with a 12-week course in MET and MBRP
  Interventions: Drug: CI-581a; Behavioral: Motivational Enhancement Therapy (MET); Behavioral: Mindfulness Based Relapse Prevention
- CI-581b+MET+MBRP (Active Comparator): Administration of CI-581b at 0.025 mg/kg during weeks 1 and 5 combined with a 12-week course in MET and MBRP
  Interventions: Drug: CI-581b; Behavioral: Motivational Enhancement Therapy (MET); Behavioral: Mindfulness Based Relapse Prevention

INTERVENTIONS:
Drug: CI-581a — Medication infusion intravenously over 1 hour.
  Arms: CI-581a+MET+MBRP
Drug: CI-581b — Medication infusion intravenously over 1 hour.
  Arms: CI-581b+MET+MBRP
Behavioral: Motivational Enhancement Therapy (MET) — Manualized one on one therapy aimed at mobilizing motivation for change and for goals.
Behavioral: Mindfulness Based Relapse Prevention — Manualized one on one therapy aimed at mindfulness-based behavioral modification and the cultivation of relapse prevention skils.

SUMMARY:
Changes in the communication of glutamate from one brain structure to another are important in the development of therapy for cocaine use disorders. Our preliminary investigations suggest that drugs that affect glutamate exchange may be effective at promoting and maintaining individuals' abstinence from cocaine. The purpose of this randomized, double-blind, controlled trial is to test various glutamate modulators in conjunction with motivational enhancement therapy (MET) and mindfulness based relapse prevention (MBRP) for cocaine use disorders.

DETAILED DESCRIPTION:
Alterations in the transmission between neurons of a neurotransmitter called glutamate are an important target of pharmacotherapy for cocaine use disorders (CUDs). Preliminary investigations suggest that glutamate modulation may be effective at promoting and maintaining abstinence and that it promotes motivation to quit, reduces craving, reduces cocaine self-administration and facilitates abstinence in individuals with a CUD in a series of trials.

The study team has recently developed and tested a novel design that integrates a clinical trial involving serial infusions and a behavioral treatment platform. The current trial will evaluate the effect of two sub-anesthetic infusions on abstinence rates in a relatively large sample of treatment-seeking CUD individuals who complete a 12-week double-blind, randomized, controlled trial. It will also evaluate the correlation between clinical response and brain-derived neurotrophic factor (BDNF), a peripheral biomarker relevant to glutamate modulation antidepressant response. This project aims to expand on several years of promising preliminary data to rigorously evaluate the efficacy of this innovative pharmacological intervention integrated into a behavioral treatment platform.

ELIGIBILITY:
Inclusion Criteria:

1. Meets DSM-V criteria for cocaine use disorders, with at least 1 day of use per week for three weeks over the past month
2. Physically healthy
3. No adverse reactions to study medications
4. 18-70 years of age
5. Capacity to consent and comply with study procedures
6. Seeking Treatment

Exclusion Criteria:

1. Meets DSM IV criteria for current major depression, bipolar disorder, schizophrenia, any psychotic illness, including substance-induced psychosis, and current substance-induced mood disorder with HAMD score > 12.
2. Physiological dependence on another substance, such as alcohol, opioids, or benzodiazepines, excluding caffeine and nicotine, requiring imminent medical management
3. Delirium, dementia, amnesia, cognitive disorders, or dissociative disorders
4. Current suicide risk or a history of suicide attempt within the 2 years
5. Pregnant, interested in becoming pregnant, or lactating
6. On psychotropic or other medication whose effect could be disrupted by participation in the study, such as benzodiazepines, opioids, or barbiturates
7. Recent history of significant violence
8. Heart disease as indicated by history, abnormal ECG, previous cardiac surgery.
9. Unstable physical disorders which might make participation hazardous such as hypertension (>160/90), anemia, active hepatitis or other liver disease (transaminase levels < 2-3 X the upper limit of normal will be considered acceptable), or untreated diabetes. Participants reporting HIV+ status will be asked to provide information about their current treatment, including all medications. Participants who are on the antiretroviral ritonavir (Norvir) will be excluded due to the possibility that study medications in combination with this medication may increase the risk of drug-induced hepatitis
10. Previous history of a substance use disorder with the study medications or benzodiazepine abuse and/or a history of adverse reaction/ experience with prior exposure to study medications or benzodiazepines

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2017-10-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Abstinence from Cocaine Use | from baseline to week 12

CONTACTS AND LOCATIONS:
Overall Officials: Elias Dakwar, MD, Principal Investigator — NYSPI
Locations (1):
- NYSPI, New York, New York, United States